CLINICAL TRIAL: NCT02260947
Title: A Double Blind, Double Dummy, Randomized, Placebocontrolled, 5 Period Cross-over Study To Examine The Effect of Pf-06273340 On Evoked Pain Endpoints In Healthy Volunteers Using Pregabalin And Ibuprofen As Positive Controls
Brief Title: Assessment of the Analgesic Effects of PF-06273340 in Healthy Volunteers Using Evoked Pain Endpoints
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: B5261005; 2014-003553-34 (EudraCT Number)
Record Dates: First submitted 2014-10-06; First posted 2014-10-09 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Healthy
MeSH Terms: interventions — PF-06273340; Pregabalin; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Experimental)
  Interventions: Drug: PF-06273340
- 2 (Experimental)
  Interventions: Drug: PF-06273340
- 3 (Active Comparator)
  Interventions: Drug: Pregabalin
- 4 (Active Comparator)
  Interventions: Drug: Ibuprofen
- 5 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-06273340 — PF-06273340 50 mg
  Arms: 1
Drug: PF-06273340 — PF-06273340 400 mg
  Arms: 2
Drug: Pregabalin — Pregabalin 300 mg
  Arms: 3
Drug: Ibuprofen — Ibuprofen 600 mg
  Arms: 4
Drug: Placebo — Matching Placebo
  Arms: 5

SUMMARY:
This study will examine the activity of 2 different doses of PF-06273340 on a panel of evoked pain tests carried out from 0.5 to 10 hours following oral dosing in healthy male subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects between the ages of 18 and 55 years, inclusive. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12 lead ECG or clinical laboratory tests.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).
* Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
* Subjects who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* A positive urine drug screen

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Thermal pain detection threshold | 0.5 - 4 hours
Ultra-violet light sensitized pain detection threshold | 0.5 - 4 hours
Pressure pain tolerance threshold | 0.5 - 4 hours
Electrical pain tolerance threshold | 0.5 - 4 hours
Cold pressor tolerance threshold | 0.5 - 4 hours

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | 0.5 - 10 hours
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 0.5 - 10 hours
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 0.5 - 10 hours
Electrical pain detection threshold | 0.5 - 10 hours
Electrical pain area under the visual analogue scale pain curve | 0.5 - 10 hours
Electrical pain post test visual analogue scale | 0.5 - 10 hours
Electrical pain post-cold pressor pain detection threshold | 0.5 - 10 hours
Electrical pain post cold pressor pain tolerance threshold | 0.5 - 10 hours
Electrical pain post cold pressor area under the visual analogue scale curve | 0.5 - 10 hours
Electrical pain post cold pressor post test visual analogue scale | 0.5 - 10 hours
Conditioned pain modulation response pain detection threshold | 0.5 - 10 hours
Conditioned pain modulation pain tolerance threshold | 0.5 - 10 hours
Conditioned pain modulation area under the visual analogue scale curve | 0.5 - 10 hours
Condition pain modulation post test VAS | 0.5 - 10 hours
Pressure pain detection threshold | 0.5 - 10 hours
Pressure pain area under the visual analogue scale curve | 0.5 - 10 hours
Pressure pain post test visual analogue scale | 0.5 - 10 hours
Cold pressor pain detection threshold | 0.5 - 10 hours
Cold pressor area under the visual analogue scale curve | 0.5 - 10 hours
Cold pressor post test visual analogue scale | 0.5 - 10 hours
PF-06273340 half life | 0.5 - 10 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Centre for Human Drug Research, Leiden, CL, Netherlands

REFERENCES:
- [Derived] Loudon P, Siebenga P, Gorman D, Gore K, Dua P, van Amerongen G, Hay JL, Groeneveld GJ, Butt RP. Demonstration of an anti-hyperalgesic effect of a novel pan-Trk inhibitor PF-06273340 in a battery of human evoked pain models. Br J Clin Pharmacol. 2018 Feb;84(2):301-309. doi: 10.1111/bcp.13448. Epub 2017 Nov 28. PMID 29178434